CLINICAL TRIAL: NCT03350139
Title: Evaluation of the Predictors of Clinical and Radiological Response to Gamma-Knife Radiosurgery in the Treatment of Intermediate Ventral Nucleus of the Thalamus (VIM) Thalamotomy Tremor.
Acronym: GARP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-09; ID RCB (Registry Identifier: 2017-A01249-44)
Record Dates: First submitted 2017-11-16; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Severe Disabling Tremor
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with gamma knife radiosurgery: Collection of non-genetic, chronobiological, therapeutic and co-morbidities
  Interventions: Device: gamma knife radiosurgery

INTERVENTIONS:
Device: gamma knife radiosurgery — The surgical procedure consists of a very partial radiation of the brain with a stereotactic precision performed in current practice

SUMMARY:
Gamma-Knife radiosurgery of the VIM for patients presenting with severe drug-resistant tremor is now current practice as an alternative to Deep Brain Stimulation (DBS) of the VIM.

Now, around 100 patients are treated annually in our unit (essential tremor or Parkinson tremor).

Clinical and radiological follow-up is demonstrating that 80% of these patients are presenting with a homogenous response complete or subtotal, the disappearance of the tremor mean delay of 6 months after radiosurgery. In neuroradiological responses on the MRI, is appearing roughly at the same time local contrast enhancement surrounding highty to signal no associated with clinical side effects.

In 15 to 20% of the patients, the clinical effets is not obtained and in the vast majority no MRI response or minimal MRI response is observed on images suggesting that these failures are related to specific resistance to radiosurgery of this subgroup.

In roughly 5% of the patients, at the contrary, hyper response is observe on the MRI rating clinically with side effects (hemiparesis or proprioceptive ataxia or dysarthria, hands problems….). The adverse effects are generally reversible either in whole or in part with the resorption of the perilesionnel oedema.

It would be extremely helpfull to be able to identify in advance these 2 groups of hyper and hypo respondeurs.

The capacity to identify in advance these patients at risk to hypo or hyper response would allow us to either contre-indicate radiosurgery or modify radiosurgery technicaly at the time of dose planing.

Sequently, these predictions would allow us to tailor individually mission management and information leading to improvment of the efficacy and tolerance of this kind of intervention.

The parameters suspected to be likely to influence the response are :

* genetics
* co-morbidities (diabetis, vascular…)
* Main aspect of the brain (severe atrophy, vascular, micro-infacts…)
* Chronobiological (timing during the day of the radiosurgical procedure)
* Associated medication (potential radioprotector or radiosensitizer effect of some drugs)
* Radiobiological (dose rate…)

The goal of this study is to collect all of these informations out of genetical one in the cohort of 700 patients having benefited ou will benefit from radiosurgery in the situation for essential tremor and parkinson disease. It will be test the predictive value of these parameters and the capacity to predict hyper or hypo response.

The work on the genetic material will take place in the second stage in the frame of a new different resarch project.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 20 years minimum
* Patient with absolute contraindication or relative to deep brain stimulation (DBS) of VIM.
* Patient having the Gamma Knife radiosurgery of VIM (combining clinical and paraclinical conditions).
* Patient affiliated to a social security scheme.
* Patient having understood and signed the information notice for non opposition.

Exclusion Criteria:

* Patient having a contraindication to performing a cerebral MRI (pace-maker, intracerebral metallic object etc.)
* Patient with a contraindication to radiosurgical treatment (previous treatment with cerebral radiotherapy)
* Vulnerable persons: minors, protected adults (guardianship or trusteeship) and adults unable to express their non-opposition.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe tremor (Essential Tremor type, Parkinson's disease tremor or others) responsible for significant functional impairment.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2017-10-23 (Actual); Primary Completion 2021-10-22 (Estimated); Study Completion 2021-10-22 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of tremor reduction in relation to clinical co-morbidity | 12 months
  Clinical response increases with decrease in clinical co-morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, General Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided